CLINICAL TRIAL: NCT01411943
Title: Epigenetic Factors Associated With Symptoms and Complications of Chronic Disorders
Brief Title: Epigenetics and Psychoneurologic Symptoms in Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM13194
Record Dates: First submitted 2011-08-03; First posted 2011-08-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Epigenetics; Inflammatory; Psychoneurologic Symptoms; Cognitive Dysfunction; Pain; Fatigue; Sleep Disturbance; Depression; Depressive Symptoms; Anxiety; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction; Pain; Fatigue; Parasomnias; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will be examining cytokine and c-reactive protein levels, DNA methylation, DNA repair proteins, telomere length and chromosomal instability.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study examines the relationship among epigenetic alterations and the development and persistence of psychoneurologic symptoms (cognitive dysfunction, depressive symptoms, anxiety, fatigue, sleep disturbance, and pain) in women receiving chemotherapy for early stage breast cancer. The relationship among inflammatory markers and psychoneurologic symptoms will also be explored. It is hypothesized:

1. Chemotherapy triggers inflammatory activation, which in turn leads to the acquisition of genetic alterations. These alterations result in cellular changes and are modified over time.
2. Inflammatory activation and epigenetic alterations are related to the temporal development, severity, and persistence of psychoneurologic symptoms.

DETAILED DESCRIPTION:
Advancements in breast cancer have resulted in increased survival rates; however, many women with breast cancer experience distressing symptoms. Inflammatory activation and epigenetic alterations have been associated with the etiology of cancer. To date, no investigators have considered these epigenetic processes as possible mechanisms associated with the etiology of distressing symptoms in women with breast cancer. The specific aims of this study are to examine:

1. The frequency and severity of psychoneurological (PN) symptoms (depressive symptoms, anxiety, sleep disturbances, fatigue, pain and cognitive dysfunction)and the interrelationship among PN symptoms at each time point
2. Levels of inflammation and to quantify the frequency and genome-wide location of changes in epigenetic patterns across time following chemotherapy
3. The relationship among inflammation, epigenetic changes, and the development, severity, and persistence of PN symptoms across time The study results may potentially deepen understanding regarding the biological processes underlying PN symptoms and lead to improved strategies for symptom management in women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Diagnosed with stage I to IIIa Breast Cancer
* Scheduled to receive chemotherapy

Exclusion Criteria:

* previous cancer history
* previous chemotherapy history
* dementia
* active psychosis

Ages: 21 Years to 81 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from oncology treatment clinics
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Epigenetics and psychoneurologic symptoms in women receiving chemotherapy for breast cancer | 5 years
  To examine the frequency and severity of psychoneurologic symptoms and the interrelatednessamong the symptoms, levels of inflammation, and the frequency and genome wide localization of changes in epigenetic patterns across time.

CONTACTS AND LOCATIONS:
Overall Officials: Debra E Lyon, PhD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Peninsula Cancer Institute, Newport News, Virginia
  - Virginia Commonwealth University, Richmond, Virginia